CLINICAL TRIAL: NCT04421937
Title: The Effects of Neuromuscular Electrical Stimulation on Swallowing Functions in Stroke Patients With Dysphagia: Randomized Controlled Trial
Brief Title: The Effects of Neuromuscular Electrical Stimulation on Swallowing Functions in Stroke Patients With Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Elif Tarihçi, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Istanbul University, Istanbul
Record Dates: First submitted 2020-05-16; First posted 2020-06-09 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Swallowing Disorder; Dysphagia; Stroke, Complication; Cerebrovascular Accident
Keywords: stroke; swallowing disorder; dysphagia; stroke rehabilitation; neuromuscular electrical stimulation; traditional dysphagia therapy
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Electrical Stimulation (NMES) with TDT (Experimental)
  Interventions: Device: Procedure: Neuromuscular Electrical Stimulation with TDT
- Traditional Dysphagia Therapy (TDT) (Active Comparator)
  Interventions: Behavioral: Procedure: Traditional Dysphagia Therapy (TDT)

INTERVENTIONS:
Behavioral: Procedure: Traditional Dysphagia Therapy (TDT) — Traditional dysphagia therapy includes diet modification training, teaching postural compensatory methods, training of oral motor control exercises and tongue root exercises, training of swallowing maneuvers, and practice of chin-resistance exercise, which is the exercise of opening the upper esophageal sphincter.
  Traditional Dysphagia Therapy will be applied for 45 minutes a day, 5 days a week for 3 weeks.
  Arms: Traditional Dysphagia Therapy (TDT)
Device: Procedure: Neuromuscular Electrical Stimulation with TDT — The skin to be treated will be cleaned and dried. NMES will be implemented with signals received from two channels. In the first channel, the upper electrodes will be placed horizontally just above the hyoid bone. This is the place where the cupping is felt when the finger is pressed right under the chin. In the second channel, the lower electrodes will be placed horizontally, just above the thyrohyoid muscle. This is the place where you can feel a cupping when pressed with your finger, on both sides of the apple in the larynx. The device will be set to start at the lowest power, with very short pulses of approximately 700 microseconds, at intervals of 1 second. The power will be gradually increased according to the device and the power that the patient feels vibration will be stopped. The power to be applied will not exceed 25 milliamps. NMES application and Traditional Dysphagia Therapy will be applied for 45 minutes a day, 5 days a week for 3 weeks.
  Arms: Neuromuscular Electrical Stimulation (NMES) with TDT

SUMMARY:
In our study, our aim is to evaluate the effect of neuromuscular electrical stimulation added to traditional dysphagia therapy in stroke patients with dysphagia, on functional oral intake status, dysphagia-related symptoms, quality of life, and complications related to dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* After the first week after a stroke, detecting dysphagia by using bedside water assessment test
* Lesion location is shown by MRI or CT
* Unsupported sitting balance
* The score of Mini-mental state examination test (MMSE) 20 and above
* Over 18 years old

Exclusion Criteria:

* Global aphasia or cognitive disorders that may affect the understanding of the instructions
* Patients with major medical problems that may affect participation
* Tracheostomy presence
* Previous neck surgery
* To have received radiotherapy in the head or neck area
* Presence of a cardiac pacemaker or a history of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Change in Functional Oral Intake Scale (FOIS) | before intervention, immediately after intervention, 3 months after the intervention
  Functional Oral Intake Scale (FOIS) is a scale that shows the functional oral intake of patients with dysphagia. FOIS used for evaluation is a two part scale consisting of 7 levels. It is used to show whether the individual is dependent on the feeding tube and the level of oral intake. On this scale, 7 shows the best and 1 shows the worst functional oral intake. The change in FOIS will be our primary outcome measure in our research. It has been evaluated as an appropriate tool to demonstrate the change in functional oral intake in stroke patients. It is suitable as an independent measure of functional oral intake in prospective studies of stroke-related dysphagia.

SECONDARY OUTCOMES:
Change in Eating Assessment Tool-10 (EAT-10) Score | before intervention, immediately after intervention, 3 months after the intervention
  Eating Assessment Tool-10 (EAT-10) is used to assess participants' dysphagia symptoms, symptom severity, and risk of oropharyngeal dysphagia. This scale is a scale of 10 questions that the patient himself answers, which questions the symptoms of dysphagia. The answer points for each question range from 0 (no problem) to 4 (serious problem). If EAT-10 score is ≥3, it is considered as "risk of oropharyngeal dysphagia". It is a useful tool to evaluate the severity of dysphagia symptom in the clinic, to monitor the progression and effectiveness of the disease.
Change in Swallowing-related Quality of Life (SWAL-QOL) Score | before intervention, immediately after intervention, 3 months after the intervention
  Swallowing-related quality of life scale (SWAL-QOL) is used to evaluate the effect of swallowing disorders on quality of life. It was created to evaluate the quality of life of patients with oropharyngeal dysphagia. It includes a total of 44 questions under eating disorder, eating time, eating desire, food selection, communication, anxiety, mental health, social functionality, fatigue, and sleep subgroups. Each question is evaluated with a score ranging from 1 (worst) to 5 (best). The subgroup scores of the scale and the total score of the scale can be used to assess the change in patients.
Change in Visual Analog Scale (VAS) | before intervention, immediately after intervention, 3 months after the intervention
  Patients' difficulty in swallowing will be questioned using the Visual Analogue Scale (VAS). On a scale of ten centimeters, patients will be asked to mark the appropriate level of dysphagia 0: No dysphagia, 10: Very severe dysphagia.
Change in Laryngostroboscopy Examination | before intervention, immediately after intervention
  In the Istanbul Faculty of Medicine Otorhinolaryngology Diseases Clinic, evaluations will be made by the Ear Nose Throat Specialist. Whether there is vocal cord paresis and paralysis and whether glottic patency is evaluated in the laryngostroboscopic examination.
Change in Fiberoptic Endoscopic Evaluation of Swallowing (FEES) | before intervention, immediately after intervention
  Fiberoptic endoscopic swallowing assessment will be performed by the otolaryngologist doctor before and immediately after the treatment. In the fiberoptic endoscopic swallowing assessment, the condition of the patient according to the penetration aspiration scale will be checked. Grade 1 represents the best and grade 7 the worst on the penetration aspiration scale.
Change in Voice-Related Quality of Life (V-RQOL) Score | before intervention, immediately after intervention, 3 months after the intervention
  This ten-item scale is a scale designed for adult populations with voice disorders to measure both social-emotional and physical-functional aspects of voice problems. The answer points for each question range from 1 (few problems) to 5 (serious problems). A total score change on this scale will be used to evaluate patients.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Tarihçi, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT04421937/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT04421937/ICF_001.pdf